CLINICAL TRIAL: NCT02598804
Title: Evaluation of the Effectiveness of Self Management Program on Changes in Physical Activity Level of Knee Osteoarthritis Patients in Spa Therapy
Acronym: GEET One
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Clermont Communauté (Other); Innovatherm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHU-251; 2015-A00831-48 (Registry Identifier: 2015-A00831-48)
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Knee Osteoarthritis; Physical Activity; Education; Self-management; Exercise
Keywords: Physical activity level; Knee osteoarthritis; Randomized controlled trials; Alternate month design study; Self-management; Self-care; Education and exercise in knee osteoarthritis; Education; Non pharmacological treatment
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

ARMS (2):
- Intervention group (Experimental): No single group but 2 groups :
  * Intervention group (5 educational workshop in addition to spa therapy)
  * Control group (Written information booklet in addition to spa therapy)
  Interventions: Other: 5 educational workshop
- control group (Other): No single group but 2 groups :
  * Intervention group (5 educational workshop in addition to spa therapy)
  * Control group (Written information booklet in addition to spa therapy)
  Interventions: Other: written information booklet

INTERVENTIONS:
Other: 5 educational workshop
  Arms: Intervention group
Other: written information booklet
  Arms: control group

SUMMARY:
The primary purpose is to evaluate the benefit of an education action of exercise on the level of physical activity in patients with knee osteoarthritis with the waning of a spa treatment for three weeks, three months after the start of the cure.

DETAILED DESCRIPTION:
The aim of this study is to prove the effectiveness of an educational intervention in thermal environment on physical activity level with knee osteoarthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, aged 50 to 75 years.
* Patients with knee osteoarthritis clinical criteria of the American College of Rheumatology (ACR)
* Patient affiliated to a social security scheme (beneficiary entitled)
* Patient registered spa
* Patient has given its consent in writing to

Exclusion Criteria:

-

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Level of physical activity at 3 month, with score on IPAQ Short form | at 3 months

SECONDARY OUTCOMES:
Self efficacy at 3 months with score on ASES | at 3 months
Functional status at 3 months with score on WOMAC | at 3 months
Fears and beliefs at 3 months with score on KOFBeQ | at 3 months
Pain at 3 months with score on EVA | at 3 months
Sarcopenia at 18 days | at 18 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Gay C, Guiguet-Auclair C, Pereira B, Goldstein A, Bareyre L, Coste N, Coudeyre E. Efficacy of self-management exercise program with spa therapy for behavioral management of knee osteoarthritis: research protocol for a quasi-randomized controlled trial (GEET one). BMC Complement Altern Med. 2018 Oct 16;18(1):279. doi: 10.1186/s12906-018-2339-x. PMID 30326906